CLINICAL TRIAL: NCT03937804
Title: New Approaches for Empowering Studies of Asthma in Populations of African Descent
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190092; 19-HG-0092
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-08-21

CONDITIONS: Asthma
Keywords: Trans-omics; Natural History
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- asthmatics: persons with asthma
- control: persons without asthma

SUMMARY:
Background:

Some groups of people have a high prevalence of asthma and allergic disease. Also, asthma and allergic disease are often found in several members of the same family. Researchers want to learn more about what factors might cause asthma, both genetic and environmental.

Objective:

To build a collection of information to try to find genes that cause conditions and disorders such as asthma and allergic disease.

Eligibility:

People ages 18 99 of self-identified African, African American, or African Caribbean descent who either have no history of asthma or wheeze or have a physician s diagnosis of asthma

Design:

Participants will be screened with an interview by phone or in person.

Participants will fill out a questionnaire about their general health and exposure to allergens and smoke.

Participants will have a physical exam.

Participants will have blood tests.

Participants will provide a skin cell sample. Up to two samples will be taken from the inside of the nose. A brush will be used to take the samples.

Participants will have a breathing test. They will be asked to blow forcefully 3 or more times into a lung function machine.

Participants may have their blood and skin samples sent to a lab. DNA will be extracted from the samples and tested.

Participants blood and skin samples will be stored. Samples may be used in future research studies.

DETAILED DESCRIPTION:
Asthma is a complex disease where the interplay between genetic factors and environmental exposures controls susceptibility and disease progression. In the U.S., there remains an epidemic of asthma that disproportionately affects underrepresented minorities and creates a major public health burden, especially among children. Asthmatics of African ancestry continue to have more severe asthma and more severe clinical symptoms than their non-African counterparts, but few studies have focused on this vulnerable group. The purpose of this study is to expand our previous study, the Consortium on Asthma among African-ancestry Populations in the Americas (CAAPA) to integrate multi-omic resources for asthma research in African Diaspora populations and by recruiting new participants. The protocol described herein refers to the recruitment that will take place at the NIH Clinical Center as part of the expansion of CAAPA (CAAPA2).

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals age 18 to 99 of self-identified African, African American, or African Caribbean ancestry who either have no history of asthma or wheeze (controls) or have a physician s diagnosis of asthma. This study focuses exclusively on African ancestry individuals in order to address a lack in the field of asthma research focusing on those of African ancestry despite the greater disease burden experienced by these individuals. Enrollment for the CAAPA2 study at the NIH CC will include only adults, while children will be enrolled at other CAAPA2 sites, consistent with expertise at those sites.

EXCLUSION CRITERIA:

* First degree relative of enrolled study participant (as determined through responses to a screening questionnaire to question on participation of parents, siblings, or half-siblings)
* Current and active smoker
* History of: chronic obstructive pulmonary disease, chronic obstructive airway disease, emphysema, chronic bronchitis, lung transplant, kyphoscoliosis, sarcoidosis, bronchopulmonary dysplasia, cystic fibrosis, bronchiectasis, rheumatoid arthritis, Crohn s disease, psoriasis, carcinoma of the lung, ciliary dyskinesia, lupus, or active tuberculosis
* Having any medical illnesses that would increase the risk that the participant would incur by participating in the study, interfere with the outcomes of the study, or interfere with the study procedures (evaluated using Spirometry Screener.)
* Current or previous COVID-19 infection
* Pregnant women: while study procedures are all minimal risk, the inclusion of pregnant women is not necessary to address the research questions. Additionally, pregnancy may affect some of our parameters of interest (particularly gene expression) in unpredictable ways and the size of the growing fetus may introduce mechanical challenges to optimal performance of pulmonary function tests at later stages of pregnancy. Exclusion will be based on self-report during screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African American adults with asthma and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Expand and integrate multi-omic resources for asthma research in African Diaspora populations and identify novel genetic determinants for risk of asthma in CAAPA cohorts | single assessment
  Expand and integrate multi-omic resources for asthma research in African Diaspora populations and identify novel genetic determinants for risk of asthma in CAAPA cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Charles N Rotimi, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD to be shared with CAAPA2 research team. De-identified IPD to be shared with CAAPA2 investigators. De-identified IPD will be shared with appropriate NIH-sponsored databases such as dbGAP and data underlying a publication may be shared with a journal requiring it for publication.
Supporting Information: Study Protocol
Time Frame: IPD has been shared with CAAPA2 Investigators at the time of collection. Data will be deposited in repositories and/or with journals at the time of publication.
Access Criteria: Other CAAPA2 Investigators from the Consortium may request access to de-identified data from all CAAPA2 sites (including this one) with an analysis plan (association studies or omics analyses) that is approved by the research team. Data shared with repositories will be controlled-access and require IRB approval.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-HG-0092.html